CLINICAL TRIAL: NCT05943119
Title: Phase II Study of Intensity Modulated Radiotherapy in Dose Painting for Sinus Carcinomas After Endoscopic Surgery
Acronym: SinocaRT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A02011-42
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Tumor, Solid
Keywords: IMRT; sinus; nasal; Mucosal toxicity
MeSH Terms: conditions — Neoplasms; Fistula | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: Radiotherapy in painting dose on histoscannographic mapping (Experimental)
  Interventions: Radiation: Radiotherapy in painting dose on histoscannographic mapping
- Control group: standard pan-sinus Radiotherapy (Active Comparator)
  Interventions: Radiation: Standard pan-sinusal Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy in painting dose on histoscannographic mapping — The target volumes to be delineated are as follows:
  * High-risk CTV (Clinical Target Volume), corresponding to all initially invaded areas, as identified by comparison between the operative report and the anatomo-pathological report (ideally with histo-surgical mapping).
  * Low-risk CTV, corresponding to naso-sinusal structures not initially invaded but at risk of recurrence, and located close to the high-risk target volume, including at least 5 mm around the high-risk volume and excluding non-risk areas (muscle, bone).
  Arms: Experimental group: Radiotherapy in painting dose on histoscannographic mapping
Radiation: Standard pan-sinusal Radiotherapy — The target volumes to be delineated are as follows:
  * High-risk CTV, including the entire post-operative cavity,
  * Low-risk CTV, adapted from the recommendations described by Lapeyre (Cancer/Radiotherapy 2005), and including at least 5 mm around the high-risk volume, excluding non-risk areas (muscle, bone).
  Arms: Control group: standard pan-sinus Radiotherapy

SUMMARY:
The patient is randomized to one of the following groups:

* Experimental group: Radiotherapy in painting dose on histoscannographic mapping
* Control group: standard pan-sinus radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Patient with a histologically confirmed malignant tumor of the sinuses, any histological type except melanoma, lymphoma, mesenchymal tumors (sarcoma)
* Patient treated by endoscopic sinonasal surgery with histosurgical mapping within 2 months prior to radiotherapy
* Indication for radiotherapy treatment (photontherapy or protontherapy), without neoadjuvant chemotherapy (concomitant chemotherapy is permitted)
* Signature of informed consent prior to any specific study procedure
* Subject affiliated to a social security system

Exclusion Criteria:

* Patient with not operated in place tumor
* Patient with distant metastases
* Patient treated with neoadjuvant chemotherapy
* Pregnant or breast-feeding woman or absence of contraception during genital activity
* History of any other malignant disease in the last 3 years, except basal cell skin cancer, carcinoma in situ or superficial bladder tumor. Any other solid tumor or lymphoma (without bone marrow involvement) must have been treated and show no sign of recurrence for at least 3 years.
* Simultaneous participation in another therapeutic clinical trial
* Patients deprived of their liberty, under guardianship, under curatorship, or subject to a legal protection measure, or unable to express their consent.
* Patients unable to undergo trial monitoring for geographical, social or psychopathological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of radiation-induced nasal, ocular, auditory, endocrine and cerebral mucosal toxicities | Toxicity grade ≥ 2 according to NCI-CTCAE V5.0 within 3 months of the end of IMRT.
  Proportion of patients who do not develop radiation-induced mucosal, ocular, auditory, endocrine and/or nervous system toxicity grade ≥ 2 according to NCI-CTCAE V5.0 within 3 months of the end of IMRT.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Francois Baclesse, Caen
  - CHU CAEN, Caen
  - Centre Oscar Lambret, Lille

IPD SHARING:
Plan to Share IPD: Undecided